CLINICAL TRIAL: NCT00927654
Title: Effect of Iloprost Inhalation Before and During Extracorporeal Circulation (ECC) on Perioperative Morbidity and Outcome in High Risk Cardiac Surgical Patients
Brief Title: Iloprost in High Risk Cardiac Surgical Patients
Acronym: Ilocard
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Algora (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. B. Zwissler, Director Clinic for Anesthesiology, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-002090-12
Record Dates: First submitted 2009-06-17; First posted 2009-06-25 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Pulmonary Hypertension
Keywords: Iloprost; pulmonary hypertension; cardio pulmonary morbidity; high risk cardiac surgical patients
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Iloprost; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iloprost (Experimental)
  Interventions: Drug: Iloprost (Ventavis)
- Isotonic Sodium Chloride solution 0.9 % (Placebo Comparator)
  Interventions: Drug: Isotonic Sodium Chloride solution 0.9 % (placebo)

INTERVENTIONS:
Drug: Iloprost (Ventavis) — Twice 20 µg at day 0 (total dose 40 µg) intraoperatively
  Other Names: Ventavis
  Arms: Iloprost
Drug: Isotonic Sodium Chloride solution 0.9 % (placebo) — Twice at day 0 intraoperatively
  Arms: Isotonic Sodium Chloride solution 0.9 %

SUMMARY:
In this study effects of the intra operative, prophylactic inhalation of Iloprost (Ventavis) before and during extracorporal circulation on perioperative morbidity and outcome in high risk cardiac surgical patients is investigated in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* for females of childbearing potential: negative pregnancy test
* patients, male or female, 18 to 85 years old
* elective open-heart surgery using heart-lung-machine
* patients with increased risk to suffer from perioperative right heart failure, i.e.,

  * protracted surgery: multiple valvular transplant or expected bypass time exceeding 120 min and/or
  * patients with preoperative known pulmonary hypertension and/or
  * patients with severe heart insufficiency (NYHA III or NYHA IV)

Exclusion Criteria:

* patient not able to give consent
* pregnant or nursing patients
* Anamnestic known hypersensitivity to the used drug (Ventavis) and its ingredients or to drugs with a similar chemical structure
* blood clotting disorder requiring treatment
* trauma, intracerebral bleeding or apoplexy within the last 3 months prior to surgery
* primary or secondary immune deficiency (e.g., pretreatment with steroids, cytostatics)
* systemic infection
* lung disorder with impaired gas exchange
* lung transplantation
* cardiac transplantation
* implantation of LVAD (left ventricular assist device)
* fluoride ulcus disorder
* planned surgery in deep hypothermia and cardiac arrest
* subconscious and psychiatric disordered patients
* participation in another clinical trial within the last 30 days prior to study start and up to 30 days after end of study
* previous participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Duration of post-operative artificial respiration after arrival on intensive care unit | 2-3 months

SECONDARY OUTCOMES:
90 days lethality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Zwissler, Prof.Dr.med., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (6):
- Germany (6):
  - Hospital of the university of Aachen, Aachen
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Hospital of the university of Duesseldorf, Düsseldorf
  - Hospital of the university of Frankfurt, Frankfurt
  - Hospital of the university of munich, Munich

REFERENCES:
- [Derived] Winterhalter M, Rex S, Stoppe C, Kienbaum P, Muller HH, Kaufmann I, Kuppe H, Dongas A, Zwissler B; ILOCARD Investigators. Effect of iloprost inhalation on postoperative outcome in high-risk cardiac surgical patients: a prospective randomized-controlled multicentre trial (ILOCARD). Can J Anaesth. 2019 Aug;66(8):907-920. doi: 10.1007/s12630-019-01309-8. Epub 2019 Feb 12. PMID 30756339